CLINICAL TRIAL: NCT05265546
Title: Investigating the Mechanisms of the Effects of Psilocybin on Visual Perception and Visual Representations in the Brain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-11-14799
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Perception Disorders
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Psilocybin 0-14 mg, before fMRI measurement
  Interventions: Drug: Psilocybin
- Comparator (Other): Psilocybin 0-14 mg, before fMRI measurement
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — The effects of different doses of psilocybin (0 - 14 mg) will be compared.

SUMMARY:
The long-term objective of this project is to characterize how psilocybin affects visual perception and the brain's representation of the visual environment. It is known that psilocybin alters aspects of visual perception, but the underlying brain mechanisms contributing to these effects are poorly understood. The proposed work will address these questions in a large, diverse sample of healthy human subjects by using functional magnetic resonance imaging (fMRI) to measure the brain's responses to visual stimuli. The proposed research will document which brain areas mediate the effects of psilocybin. The technique of fMRI will be employed to measure brain activity in different brain areas while subjects are performing a visual perceptual task.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥21 years of age at time of Informed Consent Form signing
2. Are able and willing to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations.
3. Are able to swallow capsules.
4. Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of the study.
5. Written informed consent obtained from and ability for subject to comply with the requirements of the study.
6. Have an identified support person and agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing.
7. Agree to inform the investigators within 48 hours of any new or changed medical conditions during the course of their study participation.

Exclusion Criteria:

1. Breastfeeding, have a positive pregnancy test at screening or at any point during the course of the study, or unwilling to practice birth control during participation in the study.
2. Have a current psychiatric disorder, general medical condition, or other problem or abnormality that, in the opinion of the study clinician or PI, could compromise safety, render them unsuitable for the study, or would make them unable to comply with study activities.
3. Have MRI contraindications (e.g., metal implants, pacemakers, claustrophobia etc.) as determined by an MRI contraindications questionnaire.
4. Uncontrolled hypertension (Systolic BP>139mmHG or Diastolic BP>89mmHG) or tachycardia (average HR>90bpm) averaged over at least two measurements.
5. Clinically significant cardiovascular disease (e.g., history of myocardial infarction or congestive heart failure); or baseline QT/QTc>500msec; or baseline QT/QTc 451-500msec with repeat QT/QTc >500msec.
6. Inadequate hepatic function as determined by total bilirubin or alkaline phosphatase >3x institutional upper limit of normal; or AST or ALT >6x institutional upper limit of normal. However, participants with Gilbert syndrome are allowed to enroll.
7. Inadequate renal function as determined by eGFR < 30 mL/min/1.73 m2 (based on the MDRD equation) or CrCl < 30 mL/min (based on the C-G equation).
8. The regular use of psychotropic medications, such as antidepressants (i.e., SSRIs, tricyclic antidepressants, and monoamine oxidase inhibitors), antipsychotics, and mood stabilizers.
9. Concomitant dosing of psilocybin with known UGT1A10 and UGT1A9 inhibitors (e.g., diclofenac and probenecid) will be avoided. [There is no exclusion criterion based on the use of medications or substances that are inhibitors or inducers of CYP450 enzymes.]
10. The use of Prohibited Medications:

    Serotonin Reuptake Inhibitors (SSRIs and SNRIs) Tricyclic Antidepressants (TCAs) Monoamine Oxidase Inhibitors (MAOIs) Atypical antidepressants (e.g., mirtazapine, trazodone, buspar) Antipsychotics/Neuroleptics (typical and atypical) Anti-epileptics or mood stabilizers (e.g., lithium, valproate) (does not include gabapentin used for non-epilepsy conditions) Efavirenz (Sustiva, in Atripla) Lorcaserin Over-the-counter supplements intended to affect mood or anxiety (e.g., 5HT-P, SAMe or St. John's Wort).

    Other drugs associated with the serotonin syndrome (e.g., ondansetron) used within 48 hours of study drug administration (70).

    Vasoactive drugs (e.g., sildenafil, sumatriptan, calcium channel blockers) used within 48 hours of study drug administration.
11. Unable to agree to the following required Lifestyle Modifications: Patients will be asked to refrain from consuming alcohol, cannabinoids, prescription analgesics/stimulants/benzodiazepines, and any recreational drugs for 48 hours before, the day of, and for 48 hours after study drug administration. Participants will be advised to consume their usual amount of coffee, tea, or other caffeine-containing beverages on the morning of their Medication Visits.
12. Have a recent history of suicidal ideation or attempted suicide that, in the opinion of the study clinician or PI, may present a risk of suicidal or self-injurious behavior.
13. Have received an investigational drug or taken a psychedelic within 30 days of the screening visit.
14. Have an allergy or intolerance to any of the materials contained in the investigational drug product.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude and pattern of fMRI cortical responses | Functional MRI recordings will begin approximately 30 minutes after oral administration of experimental or comparator arm treatment and will continue for up to two hours.
  Functional magnetic resonance imaging (fMRI) responses to visual stimuli will be recorded.

SECONDARY OUTCOMES:
Perceptual measurements | Statistical tests will be performed after all data collection is complete.
  Within-subject inferential statistical testing will be used to assess the effects of doses of psilocybin (0-14 mg) on participants' abilities to update prior expectations based on new information. Specifically, paired t-tests will be used to contrast perceptual measures collected at MRI scan sessions.
Voxelwise modeling | Modeling of fMRI data will be performed within subjects after experiment data collection is complete.
  Voxelwise modeling results will be quantified by measuring the amount of variance in fMRI responses to presentation of stimuli that is accounted for by the model in each voxel. Cross-validation using held-out data will be used to assess possible overfitting and to facilitate unbiased interpretations. Model weights associated with each parameter will be contrasted between the effects of doses of psilocybin (0-14 mg) and quantified for individual brain areas using paired t-tests and appropriate corrections for multiple comparisons.
Participant-reported Subjective Effects | Statistical tests will be performed after all data collection is complete.
  Within-subject inferential statistical testing will be used to assess the effects of doses of psilocybin (0 - 14 mg) on subjective effects. Specifically, paired t-tests and between-group effect sizes with 95% confidence intervals will be used to contrast patient-reported outcomes (MEQ-30, ChEQ, 11D-ASC and POMS-SF), corrected for multiple comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States